CLINICAL TRIAL: NCT05418400
Title: Comparative Study of Clinical Criteria of Different Resin Composite Restorations Among Lower Molars
Brief Title: Clinical Evaluation of Different Resin Composite Restorations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Basha, principal investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 732/385
Record Dates: First submitted 2022-06-05; First posted 2022-06-14 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Dental Caries
Keywords: composite resin
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bulkfill composites (Active Comparator): sonic fill 3 & PALFIQUE bulk flow bulk fill composite
  Interventions: Other: sonic fill 3 & PALFIQUE bulk flow & Neo spectra & Clear fill AP-X
- incremental composites (Active Comparator): Neo spectra & Clear fill AP-X incremental composites
  Interventions: Other: sonic fill 3 & PALFIQUE bulk flow & Neo spectra & Clear fill AP-X

INTERVENTIONS:
Other: sonic fill 3 & PALFIQUE bulk flow & Neo spectra & Clear fill AP-X — dental filling materials

SUMMARY:
Posterior resin composite is challenging esthetic restoration. Patients seek for durable, esthetic and functional restorations in molars. one of the major problems is polymerization shrinkage. Some materials were developed to overcome the polymerization shrinkage, among them bulk fill resin composite which have been developed to reduce the shrinkage stress during polymerization and offer much greater depth of cure. This is achieved by the addition of fillers such as barium aluminum silicate filler, ytterbium trifluoride and mixed oxides. Furthermore, a prepolymerized fillers have been added with silanes to reduce shrinkage stress. so, the objective of this trial is to clinical Evaluate and compare clinical performance of bulk fill VS incremental filling technique.

ELIGIBILITY:
Inclusion Criteria:

inclusion criteria of participants:

* Male gender
* Good oral hygiene
* Only Cooperative patient
* Medically free patient
* Age range 18-24

inclusion criteria of the teeth:

* Vital teeth with no periapical lesion or radiolucency.
* Prepared cavity with no undermined enamel walls.
* Functioning tooth with presence of an opposing.
* Healthy periodontium.

Exclusion Criteria:

* exclusion criteria of participants:

  * Old age patients
  * Patients have systemic disease or sever medically compromised
  * Patients with bruxism, clenching or temporomandibular joint disorder.
  * Por oral hygiene

exclusion criteria of teeth:

* Teeth with periapical lesions.
* Teeth with visible cracks.
* Teeth with mobility.
* Non-functioning tooth with no opposing tooth.
* Heavy occlusion or signs of sever attrition.
* Tooth with Periodontal affection.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-10-02 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Post operative sensitivity | along one year
  restorations will be evaluated the according to the modified United States Public Health Service (USPHS)
marginal discoloration | along one year
  restorations will be evaluated the according to the modified United States Public Health Service (USPHS)
marginal adaptation | along one year
  restorations will be evaluated the according to the modified United States Public Health Service (USPHS)
recurrent caries | along one year
  restorations will be evaluated the according to the modified United States Public Health Service (USPHS)

CONTACTS AND LOCATIONS:
Overall Officials: Nady Ebrahem Hasanin, professor, Study Chair — Faculty of dental medicine Al Azhar university
Locations (1):
- Faculty of dental medicine Al Azhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No